CLINICAL TRIAL: NCT02436187
Title: Guideline Recommended Care and Excess Mortality for Non ST-elevation Myocardial Infarction : A National Cohort Study
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Tatendashe Bernadette Dondo, Research assistant, University of Leeds
Other Study IDs: PG/13/81/30474
Record Dates: First submitted 2015-03-30; First posted 2015-05-06 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Non ST-elevation Myocardial Infarction
Keywords: NSTEMI; excess mortality; evidence-based care; MINAP
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to quantify the excess mortality associated with non-adherence to care for non ST-elevation myocardial infarction in England and Wales over the last decade.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or more
* patients hospitalised with non ST-elevation myocardial infarction

Exclusion Criteria:

* patients hospitalised with phenotypes other than non ST-elevation myocardial infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprised of 389,052 patients with non ST-elevation myocardial infarction admitted to hospital and were entered into Myocardial Ischaemia National Audit Project database between January 2003 and December 2013.
Sampling Method: Non-Probability Sample
Enrollment: 389057 (Actual)
Dates: Start 2003-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Mortality | Participants will be followed up for an expected average of 8 years 6 months

SECONDARY OUTCOMES:
Number of missed guideline recommended care opportunities | Participants will be followed up for an expected average of 8 years 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Gale, PhD, Principal Investigator — University of Leeds
Locations (1):
- University of Leeds, Leeds, United Kingdom

REFERENCES:
- [Background] Dondo TB, Hall M, Timmis AD, Gilthorpe MS, Alabas OA, Batin PD, Deanfield JE, Hemingway H, Gale CP. Excess mortality and guideline-indicated care following non-ST-elevation myocardial infarction. Eur Heart J Acute Cardiovasc Care. 2017 Aug;6(5):412-420. doi: 10.1177/2048872616647705. Epub 2016 May 3. PMID 27142174
- [Background] Dondo TB, Hall M, Timmis AD, Yan AT, Batin PD, Oliver G, Alabas OA, Norman P, Deanfield JE, Bloor K, Hemingway H, Gale CP. Geographic variation in the treatment of non-ST-segment myocardial infarction in the English National Health Service: a cohort study. BMJ Open. 2016 Jul 12;6(7):e011600. doi: 10.1136/bmjopen-2016-011600. PMID 27406646